CLINICAL TRIAL: NCT07197073
Title: Evaluation of the Antibacterial Effect of Ozonated Olive Oil, Propolis, and Chlorhexidine Mouthwashes in Pediatric Patients: A Randomized Controlled Clinical Trial
Brief Title: Antibacterial Effect of Ozonated Olive Oil, Propolis and Chlorhexidine Mouthwashes in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0937_07/2024
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Oral Hygiene; Oral Health
Keywords: Ozonated olive oil; Chlorhexidine; Antibacterial; Propolis
MeSH Terms: interventions — Propolis; Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ozonated olive oil mouthwash (Experimental)
  Interventions: Other: Ozonated olive oil
- Propolis mouthwash (Experimental)
  Interventions: Other: Propolis
- Chlorhexidine mouthwash (Active Comparator)
  Interventions: Other: Chlorhexidine

INTERVENTIONS:
Other: Ozonated olive oil — Ozonated olive oil mouthwash will be prepared by Smart Ozone Marvel using by company's ozone. Children will be instructed to use 10 ml of mouthwash for 1 minute twice daily after 1 hour after tooth brushing
  Arms: Ozonated olive oil mouthwash
Other: Propolis — Propolis mouthwash will be prepared by using 2% raw propolis, 40 ml flavouring and 0.1 gm coloring agents, 150 ml propylene glycol, and 60 gm sorbitol. Children will be instructed to use 10 ml of mouthwash for 1 minute twice daily after 1 hour after tooth brushing
  Arms: Propolis mouthwash
Other: Chlorhexidine — The patients were given 0.12% Chlorhexidine. Children will be instructed to use 10 ml of mouthwash for 1 minute twice daily after 1 hour after tooth brushing
  Arms: Chlorhexidine mouthwash

SUMMARY:
Streptococcus mutans and Lactobacillus acidophilus are the most common cariogenic microorganisms. Chlorhexidine has been the most widely used antibacterial mouthwash in dentistry. On the other hand, few studies have reported the antibacterial potential of Propolis and Ozonated olive oil as antibacterial agents that can be used as alternatives to Chlorhexidine. This study aims to evaluate and compare the antibacterial effect of Ozonated olive oil, Propolis, and Chlorhexidine on S. mutans and L. acidophilus count in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* High caries risk patients, according to AAPD guidelines, with visible caries or radiographic penetration into dentin, white spots on smooth surfaces, or recent restorations or missing teeth due to caries.
* Cooperative children according to Frankl's rating (score 3 & 4)

Exclusion Criteria:

* Children with any medical illness or oral infection or those who received any type of antibiotic treatment or mouthwash for two weeks before or during the study were excluded

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Change in microbial count | Baseline and after 14 days of treatment
  Total bacterial count before and after the intervention was detected. plaque samples were dispersed by vortexing for 30 seconds then 10 fold serially diluted using sterile saline.
Change in plaque accumulation | Baseline and after 14 days of treatment
  The plaque accumulation was scored for each tooth on its four surfaces.The number of positively scored surfaces is divided by the total number of tooth surfaces evaluated and the result is multiplied by 100 to express the index as a percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Pediatric dentistry, Faculty of dentistry, Alexandria University, Egypt, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No